CLINICAL TRIAL: NCT03823365
Title: Immune Reconstitution With Blinatumomab Expanded T-cells (BET) After First-line Treatment With Fludarabine-Cyclophosphamide-Rituximab or Bendamustine-Rituximab in CD20+ Indolent Non-Hodgkin Lymphomas/Chronic Lymphocytic Leukemia: a Phase I Study
Brief Title: Blinatumomab Expanded T-cells (BET) in Indolent Non-Hodgkin Lymphomas/Chronic Lymphocytic Leukemia
Acronym: BET2017
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Rambaldi Alessandro, Head Hematology and Bone Marrow Transplant, A.O. Ospedale Papa Giovanni XXIII
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Nr 2018-000086-36
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Indolent Non-Hodgkin Lymphomas/Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: CD20+ Indolent Non-Hodgkin Lymphomas/Chronic Lymphocytic Leukemia Patients After First-line Treatment with Fludarabine-Cyclophosphamide-Rituximab or Bendamustine-Rituximab.
Masking Description: This study is a phase I open-label, single center study. The patient population will consist of adults diagnosed with indolent non-Hodgkin lymphomas (iNHL) or chronic lymphocytic leukemia (CLL) in need of first line treatment consisting of either FCR or BR as per investigator assessment. Chemotherapy treatment will consist of a minimum of 4 to a maximum of 6 cycles of standard FCR or BR.Patients will be enrolled in the study after the last planned cycle of chemo-immunotherapy and, if eligibility criteria are met, BET dose level will be assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indolent NHL or CLL patients (Experimental): Adults diagnosed with indolent non-Hodgkin lymphomas (iNHL) or chronic lymphocytic leukemia (CLL) in need of first line treatment consisting of either FCR or BR as per investigator assessment
  Interventions: Biological: Blinatumomab Expanded T-cells (BET)

INTERVENTIONS:
Biological: Blinatumomab Expanded T-cells (BET) — Two to five days after the last chemotherapy infusion, BET will be administered. An accelerated titration dose escalation design will be used. During dose escalation, up to four dose levels (see table) will be evaluated or until (Maximum Tolerated Dose) MTD is reached.
  Dose level BET dose(Counted on CD3+ cells)
  1. (starting dose) 3.0 x 109
  2. 6.0 x 109
  3. 9.0 x 109
  4. 12.0 x 109

SUMMARY:
Non-Hodgkin CD20 + Indolent Lymphoma (iNHL) and Chronic Lymphatic Leukemia (CLL) are the most frequent neoplasms of B lymphocytes. They include various histologies (follicular NHL, marginal zone NHL and Lymphocytic NHL/ CLL) characterized by a chronic course and prolonged survival, but while patients with a limited disease could be cured, those with advanced disease or relapsed after localized radiation therapy are generally considered untreatable through standard treatments. The options for first-line therapy include the use of the FCR scheme, based on Fludarabine, Cyclophosphamide and Rituximab or the BR, with Bendamustine and Rituximab. Despite good results, treatment with these two regimens (FCR or BR) is associated with severe immunosuppression which worsens the immunological dysfunction already present at diagnosis in several patients. It has been shown previously that the adoptive transfer of ex vivo anti-CD3/CD28 co-stimulated autologous T cells can successfully accelerate a robust early recovery of T cells after autologous transplantation in multiple myeloma. These CD3/CD28 expanded T cells cannot however be used in NHLi and CLL due to the presence of contaminating tumor cells in the preparation. Polyclonal T cells can also be expanded in vitro in presence of Blinatumomab and recombinant human IL2 (rhIL2) and have been called BET (Blinatumomab-expanded T cells). They are a product of Advanced Therapeutic Medicinal Product (ATMP) composed of polyclonal CD8 and CD4 T cells that are still functional and devoid of contaminating CD19+ neoplastic cells. Based on these data, it was hypothesized that infusion of BET in patients with iNHL/CLL, after the first treatment line (with FCR or BR), could induce adequate immunological recovery.

DETAILED DESCRIPTION:
* Indolent non-Hodgkin lymphomas (iNHL) and chronic lymphocytic leukemia (CLL) are among the most frequent B-cell neoplasms. They include different histologies (i.e. follicular NHL, marginal zone NHL and lymphocytic NHL/CLL) characterized by chronic course and prolonged survival. While some patients with limited stage disease may be cured, those presenting with advance stage or relapsing after local radiotherapy are generally considered not curable with standard treatments.
* First-line treatment of CLL/LL is currently based on the biologic profile of the disease. Excluding high risk patients harboring the del(17p) and/or TP53 mutations, first line chemoimmunotherapy options includes the use of either fludarabine, cyclophosphamide and rituximab (FCR) or BR. Despite the good results, treatment with FCR or BR regimens is associated with severe immunosuppression that worsens the immune dysfunctions already present at diagnosis in several patients. In the CLL phase III trial, high frequency of grade 3/4 infections was reported in FCR and BR, being observed in 39% and 25% of the patients, respectively. In iNHL, infections have been observed in 37-55% of the patients treated with BR, with grade 3/4 events in 7-12% of the cases.
* Blinatumomab-expanded T cells (BET) are an Advanced Therapeutic Medicinal Product (ATMP) composed of autologous polyclonal activated T cells expanded in vitro using blinatumomab and rhIL-2, to be used for somatic cell therapy in an autologous setting. Indeed the investigators have developed a method using blinatumomab and rhIL2 to expand and activate ex vivo the T lymphocytes present in the peripheral blood from CLL and iNHL patients, while at the same time eliminating contaminating CD19+ neoplastic cells. The resulting polyclonal T cells can be used for immuno-reconstitution purposes. The Cell Factory "Centro di Terapia Cellulare G. Lanzani" showed the functionality of BET in a mouse B-cell NHL xenograft model. Upon in vivo inoculation, BET retain functional activity: upon engagement with blinatumomab in vivo, BET were able to efficiently kill the B-cell NHL cells. Importantly, BET did not showed any toxicity in animals, even at high doses and in presence of blinatumomab.
* About clinical experience, it has been previously shown that adoptive transfer of ex vivo (anti-CD3/anti-CD28) co-stimulated autologous T cells can successfully accelerate a robust T-cell recovery early after autologous transplant for multiple myeloma. However, the invariable presence of clonal disease in cell product of iNHL/CLL patients hampered this possibility up to now. In contrast BET cell expansion leads to lysis of contaminating neoplastic cells. BET can therefore be expanded from CLL patients peripheral blood in GMP (Good Manufacturing Practice) conditions for adoptive therapy. Starting from only 10 mL of peripheral blood, a mean 5.15x108 CD3+ cells can be expanded in 3 weeks with a rapid clearance of CLL contamination. The resulting blinatumomab-expanded T cells (BET) were polyclonal CD4+ and CD8+ T cells and mostly effector and central memory cells. They showed a normalized expression of the synapse inhibitors CD272 and CD279 compared with starting T cells and were functionally active, showing cytotoxicity against CD19+ targets in presence of Blinatumomab in vitro and in vivo.
* On the basis of these data the investigators hypothesize that BET infusion after first-line treatment of iNHL/CLL with either FCR or BR could lead to an adequate immune recovery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients 18 years or older 2. Confirmed diagnosis of the following CD20+ iNHL or CLL according to (World Health Organization ) WHO criteria:

  * Follicular NHL
  * Marginal zone NHL (splenic, extranodal or nodal)
  * Lymphocytic lymphoma/CLL without del(17p) or TP53 mutations 3. No previous chemotherapy. Previous radiotherapy for localized disease is admitted 4. Requirement for treatment:
  * For CLL, active disease is defined as meeting at least one of the International Workshop on CLL guidelines (Hallek et al., 2008)
  * For iNHL, active disease is defined as meeting at least one of the Groupe d'Etudes des Lymphomes Folliculaires (GELF) criteria (Brice et al., 1997) 5. Indication to treatment with either fludarabine, cyclophosphamide and rituximab or bendamustine and rituximab 6. Presence of peripheral blood clone ≥10% of total lymphocytes (with absolute lymphocyte count >800 x106/L) at study entrance 7. Written informed consent prior to any study procedures being performed

Additional inclusion criteria to be met at study entry (i.e. before BET infusion):

8. Achieving at least a partial response after three chemo-immunotherapy cycles 9. Absence of any serious therapy-related complications that might affect interpretation of the results of the study or render the subject at high risk from treatment complications 10. Production of adequate BET numbers (counted on CD3+ cells: ≥0.5 x 109) 11. For female patients:

1. being postmenopausal for at least 1 year before the screening visit, OR
2. being surgically sterile, OR
3. if they are of childbearing potential, must agree to practice highly effective method of contraception and one additional effective (barrier) method from the time of signing the informed consent until the end of study. Highly effective method of contraception includes: (i) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal; (ii) progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable (intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence) OR
4. must agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject from the time of signing the informed consent until the end of study. [Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.]

For male patients, even if surgically sterilized (i.e., status postvasectomy):

1. with female partners of childbearing potential: must agree to practice barrier contraception (condom with or without spermicide) from the time of signing the informed consent until the end of study and his female partner must agree to practice method of contraception including one of the following: estrogen and progestogen containing hormonal contraception; inhibition of ovulation: oral, intravaginal, transdermal; progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable (intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion) from the time of signing the informed consent until the end of study.
2. must agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject from the time of signing the informed consent until the end of study. [Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.]
3. must agree to refrain from donating sperm

Exclusion Criteria:

1. ECOG (Eastern Cooperative Oncology Group) Performance Status >2
2. Active central nervous system (CNS) disease
3. Calculated creatinine clearance (by Cockroft-Gault) of < 50 ml/min or serum creatinine > 1.5x ULN (Upper Limit of Normal )
4. Concomitant or previous diagnosis of autoimmune hemolytic anemia or thrombocytopenia
5. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring the sole hormone replacement are allowed to participate. Psoriasis requiring systemic treatment, or conditions expected to recur at the presence of an external trigger are excluded.
6. Known infection with human immunodeficiency virus (HIV) or treponema
7. Active hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infections
8. Any suspected or known active infection
9. History of other diseases, metabolic dysfunctions, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications
10. Residual CD19+ B cells in BET final cell product ≥0.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Number of grade 3 or 4 adverse events (AE) possibly related to therapy | The period of observation is during 14 days after BET infusion
  Description and grading of all adverse events will be based on the NCI -CTCAE v4.03 and MedDra code (current version).

SECONDARY OUTCOMES:
Number of Adverse event (AE) and laboratory abnormalities. | From date of study start up to 180 days after BET infusion
  Number, causality and intensity of all adverse events will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.03 and MedDRA code (current version).
Evaluation of Optimal Biological Dose (ODB) of BET cells | +90 days after infusion
  OBD of BET will be defined as the absolute number of BET cell that will allow a CD3+ count of > 600 x106/L at +90 days after infusion in at least 70% of the patients.
Evaluation of general Immune Reconstitution after BET infusion | at +0 (4 hours), +30, +90 and +180 days after infusion
  Absolute numbers of B, T, and NK cells reconstitution and its correlation with BET cell infused and its composition (in terms of T-cell subsets and NK cells)
Evaluation of ex vivo transfer of anti-viral immunity | at +0 (4 hours), +30, +90 and +180 days after infusion
  Ex vivo transfer of anti-viral immunity in terms of tetramer-based quantification of CMV-specific CD8+ T lymphocytes (this will be done only for CMV positive patients for whom CMV specific tetramers stain positive in starting peripheral blood or BET).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — ASST - Papa Giovanni XXIII
Locations (1):
- ASST - Papa Giovanni XXIII, Bergamo, Italy

REFERENCES:
- [Background] Ardeshna KM, Smith P, Norton A, Hancock BW, Hoskin PJ, MacLennan KA, Marcus RE, Jelliffe A, Vaughan G, Hudson, Linch DC; British National Lymphoma Investigation. Long-term effect of a watch and wait policy versus immediate systemic treatment for asymptomatic advanced-stage non-Hodgkin lymphoma: a randomised controlled trial. Lancet. 2003 Aug 16;362(9383):516-22. doi: 10.1016/s0140-6736(03)14110-4. PMID 12932382
- [Background] Berdeja JG, Hess A, Lucas DM, O'Donnell P, Ambinder RF, Diehl LF, Carter-Brookins D, Newton S, Flinn IW. Systemic interleukin-2 and adoptive transfer of lymphokine-activated killer cells improves antibody-dependent cellular cytotoxicity in patients with relapsed B-cell lymphoma treated with rituximab. Clin Cancer Res. 2007 Apr 15;13(8):2392-9. doi: 10.1158/1078-0432.CCR-06-1860. PMID 17438098
- [Background] Bomberger C, Singh-Jairam M, Rodey G, Guerriero A, Yeager AM, Fleming WH, Holland HK, Waller EK. Lymphoid reconstitution after autologous PBSC transplantation with FACS-sorted CD34+ hematopoietic progenitors. Blood. 1998 Apr 1;91(7):2588-600. PMID 9516161
- [Background] Brice P, Bastion Y, Lepage E, Brousse N, Haioun C, Moreau P, Straetmans N, Tilly H, Tabah I, Solal-Celigny P. Comparison in low-tumor-burden follicular lymphomas between an initial no-treatment policy, prednimustine, or interferon alfa: a randomized study from the Groupe d'Etude des Lymphomes Folliculaires. Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 1997 Mar;15(3):1110-7. doi: 10.1200/JCO.1997.15.3.1110. PMID 9060552
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Chemotherapeutic options in chronic lymphocytic leukemia: a meta-analysis of the randomized trials. CLL Trialists' Collaborative Group. J Natl Cancer Inst. 1999 May 19;91(10):861-8. doi: 10.1093/jnci/91.10.861. PMID 10340906
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Darwish M, Bond M, Hellriegel E, Robertson P Jr, Chovan JP. Pharmacokinetic and pharmacodynamic profile of bendamustine and its metabolites. Cancer Chemother Pharmacol. 2015 Jun;75(6):1143-54. doi: 10.1007/s00280-015-2727-6. Epub 2015 Apr 1. PMID 25829094
- [Background] Grupp SA, Kalos M, Barrett D, Aplenc R, Porter DL, Rheingold SR, Teachey DT, Chew A, Hauck B, Wright JF, Milone MC, Levine BL, June CH. Chimeric antigen receptor-modified T cells for acute lymphoid leukemia. N Engl J Med. 2013 Apr 18;368(16):1509-1518. doi: 10.1056/NEJMoa1215134. Epub 2013 Mar 25. PMID 23527958
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Introna M, Borleri G, Conti E, Franceschetti M, Barbui AM, Broady R, Dander E, Gaipa G, D'Amico G, Biagi E, Parma M, Pogliani EM, Spinelli O, Baronciani D, Grassi A, Golay J, Barbui T, Biondi A, Rambaldi A. Repeated infusions of donor-derived cytokine-induced killer cells in patients relapsing after allogeneic stem cell transplantation: a phase I study. Haematologica. 2007 Jul;92(7):952-9. doi: 10.3324/haematol.11132. PMID 17606446
- [Background] Introna M, Pievani A, Borleri G, Capelli C, Algarotti A, Mico C, Grassi A, Oldani E, Golay J, Rambaldi A. Feasibility and safety of adoptive immunotherapy with CIK cells after cord blood transplantation. Biol Blood Marrow Transplant. 2010 Nov;16(11):1603-7. doi: 10.1016/j.bbmt.2010.05.015. Epub 2010 Jun 1. PMID 20685246
- [Background] Kalamasz D, Long SA, Taniguchi R, Buckner JH, Berenson RJ, Bonyhadi M. Optimization of human T-cell expansion ex vivo using magnetic beads conjugated with anti-CD3 and Anti-CD28 antibodies. J Immunother. 2004 Sep-Oct;27(5):405-18. doi: 10.1097/00002371-200409000-00010. PMID 15314550
- [Background] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Background] Levine BL, Bernstein WB, Connors M, Craighead N, Lindsten T, Thompson CB, June CH. Effects of CD28 costimulation on long-term proliferation of CD4+ T cells in the absence of exogenous feeder cells. J Immunol. 1997 Dec 15;159(12):5921-30. PMID 9550389
- [Background] Levine BL, Cotte J, Small CC, Carroll RG, Riley JL, Bernstein WB, Van Epps DE, Hardwick RA, June CH. Large-scale production of CD4+ T cells from HIV-1-infected donors after CD3/CD28 costimulation. J Hematother. 1998 Oct;7(5):437-48. doi: 10.1089/scd.1.1998.7.437. PMID 9829318
- [Background] Loffler A, Gruen M, Wuchter C, Schriever F, Kufer P, Dreier T, Hanakam F, Baeuerle PA, Bommert K, Karawajew L, Dorken B, Bargou RC. Efficient elimination of chronic lymphocytic leukaemia B cells by autologous T cells with a bispecific anti-CD19/anti-CD3 single-chain antibody construct. Leukemia. 2003 May;17(5):900-9. doi: 10.1038/sj.leu.2402890. PMID 12750704
- [Background] Long-Boyle JR, Green KG, Brunstein CG, Cao Q, Rogosheske J, Weisdorf DJ, Miller JS, Wagner JE, McGlave PB, Jacobson PA. High fludarabine exposure and relationship with treatment-related mortality after nonmyeloablative hematopoietic cell transplantation. Bone Marrow Transplant. 2011 Jan;46(1):20-6. doi: 10.1038/bmt.2010.53. Epub 2010 Apr 12. PMID 20383215
- [Background] Mackall CL. T-cell immunodeficiency following cytotoxic antineoplastic therapy: a review. Oncologist. 1999;4(5):370-8. PMID 10551553
- [Background] Maus MV, Thomas AK, Leonard DG, Allman D, Addya K, Schlienger K, Riley JL, June CH. Ex vivo expansion of polyclonal and antigen-specific cytotoxic T lymphocytes by artificial APCs expressing ligands for the T-cell receptor, CD28 and 4-1BB. Nat Biotechnol. 2002 Feb;20(2):143-8. doi: 10.1038/nbt0202-143. PMID 11821859
- [Background] Nagorsen D, Baeuerle PA. Immunomodulatory therapy of cancer with T cell-engaging BiTE antibody blinatumomab. Exp Cell Res. 2011 May 15;317(9):1255-60. doi: 10.1016/j.yexcr.2011.03.010. Epub 2011 Mar 16. PMID 21419116
- [Background] Rapoport AP, Stadtmauer EA, Aqui N, Badros A, Cotte J, Chrisley L, Veloso E, Zheng Z, Westphal S, Mair R, Chi N, Ratterree B, Pochran MF, Natt S, Hinkle J, Sickles C, Sohal A, Ruehle K, Lynch C, Zhang L, Porter DL, Luger S, Guo C, Fang HB, Blackwelder W, Hankey K, Mann D, Edelman R, Frasch C, Levine BL, Cross A, June CH. Restoration of immunity in lymphopenic individuals with cancer by vaccination and adoptive T-cell transfer. Nat Med. 2005 Nov;11(11):1230-7. doi: 10.1038/nm1310. Epub 2005 Oct 16. PMID 16227990
- [Background] Rapoport AP, Stadtmauer EA, Aqui N, Vogl D, Chew A, Fang HB, Janofsky S, Yager K, Veloso E, Zheng Z, Milliron T, Westphal S, Cotte J, Huynh H, Cannon A, Yanovich S, Akpek G, Tan M, Virts K, Ruehle K, Harris C, Philip S, Vonderheide RH, Levine BL, June CH. Rapid immune recovery and graft-versus-host disease-like engraftment syndrome following adoptive transfer of Costimulated autologous T cells. Clin Cancer Res. 2009 Jul 1;15(13):4499-507. doi: 10.1158/1078-0432.CCR-09-0418. Epub 2009 Jun 9. PMID 19509133
- [Background] Robak T, Lech-Maranda E, Korycka A, Robak E. Purine nucleoside analogs as immunosuppressive and antineoplastic agents: mechanism of action and clinical activity. Curr Med Chem. 2006;13(26):3165-89. doi: 10.2174/092986706778742918. PMID 17168705
- [Background] Rummel MJ, Niederle N, Maschmeyer G, Banat GA, von Grunhagen U, Losem C, Kofahl-Krause D, Heil G, Welslau M, Balser C, Kaiser U, Weidmann E, Durk H, Ballo H, Stauch M, Roller F, Barth J, Hoelzer D, Hinke A, Brugger W; Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. Lancet. 2013 Apr 6;381(9873):1203-10. doi: 10.1016/S0140-6736(12)61763-2. Epub 2013 Feb 20. PMID 23433739
- [Background] Saito H, Maruyama D, Maeshima AM, Makita S, Kitahara H, Miyamoto K, Fukuhara S, Munakata W, Suzuki T, Kobayashi Y, Taniguchi H, Tobinai K. Prolonged lymphocytopenia after bendamustine therapy in patients with relapsed or refractory indolent B-cell and mantle cell lymphoma. Blood Cancer J. 2015 Oct 23;5(10):e362. doi: 10.1038/bcj.2015.86. No abstract available. PMID 26495859
- [Background] Solal-Celigny P, Bellei M, Marcheselli L, Pesce EA, Pileri S, McLaughlin P, Luminari S, Pro B, Montoto S, Ferreri AJ, Deconinck E, Milpied N, Gordon LI, Federico M. Watchful waiting in low-tumor burden follicular lymphoma in the rituximab era: results of an F2-study database. J Clin Oncol. 2012 Nov 1;30(31):3848-53. doi: 10.1200/JCO.2010.33.4474. Epub 2012 Sep 24. PMID 23008294
- [Background] Stadtmauer EA, Vogl DT, Luning Prak E, Boyer J, Aqui NA, Rapoport AP, McDonald KR, Hou X, Murphy H, Bhagat R, Mangan PA, Chew A, Veloso EA, Levine BL, Vonderheide RH, Jawad AF, June CH, Sullivan KE. Transfer of influenza vaccine-primed costimulated autologous T cells after stem cell transplantation for multiple myeloma leads to reconstitution of influenza immunity: results of a randomized clinical trial. Blood. 2011 Jan 6;117(1):63-71. doi: 10.1182/blood-2010-07-296822. Epub 2010 Sep 23. PMID 20864577
- [Background] Swerdlow SH, Campo E, Pileri SA, Harris NL, Stein H, Siebert R, Advani R, Ghielmini M, Salles GA, Zelenetz AD, Jaffe ES. The 2016 revision of the World Health Organization classification of lymphoid neoplasms. Blood. 2016 May 19;127(20):2375-90. doi: 10.1182/blood-2016-01-643569. Epub 2016 Mar 15. PMID 26980727
- [Background] Wong R, Pepper C, Brennan P, Nagorsen D, Man S, Fegan C. Blinatumomab induces autologous T-cell killing of chronic lymphocytic leukemia cells. Haematologica. 2013 Dec;98(12):1930-8. doi: 10.3324/haematol.2012.082248. Epub 2013 Jun 28. PMID 23812940
- [Background] Ysebaert L, Gross E, Kuhlein E, Blanc A, Corre J, Fournie JJ, Laurent G, Quillet-Mary A. Immune recovery after fludarabine-cyclophosphamide-rituximab treatment in B-chronic lymphocytic leukemia: implication for maintenance immunotherapy. Leukemia. 2010 Jul;24(7):1310-6. doi: 10.1038/leu.2010.89. Epub 2010 May 13. PMID 20463751